CLINICAL TRIAL: NCT05276648
Title: Efficacy of Erector Spinae Plane Block on Postoperative Delirium in Patients Undergoing Lumbar Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, BULUT POLAT, DR, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/05
Record Dates: First submitted 2022-01-31; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP BLOCK (Experimental): erector spina plane block applied
  Interventions: Diagnostic Test: CAM ICU test; Diagnostic Test: MOCA test; Diagnostic Test: brief pain test; Diagnostic Test: VAS scale
- no ESP BLOCK (Active Comparator): those who did not apply erector spina plan block
  Interventions: Diagnostic Test: CAM ICU test; Diagnostic Test: MOCA test; Diagnostic Test: brief pain test; Diagnostic Test: VAS scale

INTERVENTIONS:
Diagnostic Test: CAM ICU test — CAM ICU for delirium
Diagnostic Test: MOCA test — MOCA for cognitif disfonction
Diagnostic Test: brief pain test — BRİEF PAİN for chronic pain
Diagnostic Test: VAS scale — VAS scale for acute pain

SUMMARY:
Lumbar vertebra surgery is one of the most common surgical procedures.Delirium is common in geriatric patients after lumbar spinae surgery.postoperative delirium usually occurs in the early postoperative period and delays patient mobilization and thus lengthens hospital stay.

The aim of this study was to investigate the effect of this field block on postoperative delirium in patients undergoing ESP with lomber vertebra surgery and with ultrasound guidance for postoperative analgesia.

DETAILED DESCRIPTION:
Postoperative delirium (PD) and postoperative cognitive dysfunction (POCD) are extremely common in geriatric surgical patients. After elective major joint replacement or other types of major surgery, about 5% to 15% of elders develop delirium and 25% to 40% and 12% to 15% developearly or late POCD. PDand POCD are associated with prolonged length of stay, discharge to a place other than home and higher 1 year mortality. In addition, delirium is associated with an accelerated trajectory of cognitive decline to dementia (1). The etiologies of both PD and POCD remain unknown. Controversy exists over whether delirium is a marker or risk factor for subsequent persistent cognitive impairment . The PD is an acute impairment of cognitive and or spatial/temporal perception,that can be diagnosed at the bedside with dedicated diagnostic tools. It has an acute onset and a fluctuating course, and therefore can be missed if not systematically tested. It is defined by three principal characteristics: altered consciousness; changes in cognitive abilities; recent and rapid onset . The POCD affects global cognitive functions for several months/years after surgery and anesthesia, diagnosis requires detailed neuropsychological testing.

Surgical interventions have been associated with severe pain and discomfort in the immediate perioperative period. Surgical anesthesia and the perioperative analgesic regimen aim toward complete intra-operative amnesia, profound analgesia, effective control of autonomic responses and rapid emergence. However, anesthesia, analgesia and sedation all utilize medications that might be implicated in the development of central nervous system (CNS) dysfunction. Elderly patients are more sensitive to the CNS effects of barbiturates, inhalationalanesthetics, benzodiazepines and opioids. Some medications frequently associated with delirium with or without POCD include opioids, anxiolytics, antidepressants, and corticosteroids.

There are studies regarding the effect of erektor spina field block on postoperative pain in vertebra surgery.The investigators will compare the effect on postoperative delirium of patients who underwent erector spina plane block after spinal surgery with those who did not.

ELIGIBILITY:
Inclusion Criteria:

1. 60 and older
2. ASA Physical Status 1-3;
3. Scheduled for elective hip surgery under spinal anesthesia
4. MMSE ≥ 20 (to exclude dementia)

Exclusion Criteria:

1. Severe visual or auditory disorder/handicaps
2. Bipolar disorder
3. major depression
4. schizophrenia
5. Alzheimer
6. Dementia
7. ASA physical status IV or V

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effect of postoperative delirium (determined by CAM ICU test) in patients who underwent erector spina block after spinal surgery and those who did not. | Change from baseline postoperative delirium at five days
  CAM ICU IS THE TEST USED TO MEASURE DELIRIUM

SECONDARY OUTCOMES:
postoperative chronic pain assessment.we will use brief pain scoring | 3 month later (one time)
  brief pain scoring is the test used to measure chronic pain
postoperative cognitive dysfunction assessment.we will use montreal cognitive assesment test | 3 month later (one time)
  montreal cognitive assesment is the test used to measure postoperative cognitive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Sari öztürk, Study Director — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No